CLINICAL TRIAL: NCT00607425
Title: Saliva mRNA Expression Profiling for Early Stage Non-Small Cell Lung Cancer Screening
Acronym: SPIT-LC
Status: Terminated | Type: Observational
Why Stopped: Change in isolation method
Sponsor: Scottsdale Healthcare (Other)
Collaborators: University of California, Los Angeles (Other); University of Colorado, Denver (Other); US Department of Veterans Affairs (U.S. Federal Agency); University of Kansas (Other)
Responsible Party: Glen J. Weiss, MD, TGen Clinical Research Services at Scottsdale Healthcare
Other Study IDs: 2007-094; IASLC
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; screening; saliva; gene expression; healthy control subject
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Non-small cell lung cancer patients
- 2: Healthy control subjects

SUMMARY:
This is a pilot study to test the feasibility of using gene expression from saliva to identify patients with early-stage non-small cell lung cancer (NSCLC).

The primary objective of this study is to compare gene expression profiles from saliva from healthy controls and patients with early-stage non-small cell lung cancer.

To be eligible, patients with non-small cell lung cancer, must not yet have received treatment for their cancer (surgical removal, chemotherapy, or radiation therapy). Health control participants may participate if they meet eligibility criteria listed below.

Eligible enrollees will be asked to submit a one time saliva sample and complete a study questionaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with untreated stage I-II NSCLC OR Healthy control subjects: with a > 20 pack year history of cigarette smoking OR Never smokers (defined as less than 100 cigarettes over subject's lifetime)

   * The investigators recognize that pathologic confirmation is not always available prior to surgical resection of a lung mass. To account for this, subjects with a suspicious lung mass concerning for lung cancer, can be enrolled on this trial, and submit a saliva sample prior to surgical resection (ideally within 45 days of planned surgery).
2. Adults age 40-79
3. Ability to understand the investigational nature of the study and sign the informed consent in accordance with institutional and FDA guidelines

Exclusion Criteria:

1. No active pulmonary infection, i.e. bronchitis or pneumonia for 6 months
2. No use of steroid inhalers for > 6 months
3. No other prior malignancy is allowed except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancers from which the patient has been disease-free for 5 years

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Untreated, clinical stage I and II non-small cell lung cancer (NSCLC) patients and matching healthy control subjects will be recruited to participate in this study.
  Untreated patients have not yet had either complete surgical removal of their lung cancer, any chemotherapy, or any radiation therapy to treat their lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen J Weiss, MD, Principal Investigator — TGen Clinical Research Services at Scottsdale Healthcare